CLINICAL TRIAL: NCT00458744
Title: A Phase I Study Of Talotrexin (PT-523) In Children And Adolescents With Recurrent Solid Tumors Or Recurrent/Refractory Leukemias
Brief Title: Talotrexin in Treating Young Patients With Recurrent Solid Tumors or Leukemia That is Recurrent or Does Not Respond to Treatment
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study withdrawn because of toxicity reported on the adult phase 1 trial.
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ADVL0613; COG-ADVL0613 (Other: Children's Oncology Group); CDR0000538359 (Other: Clinical Trials.gov)
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Brain and Central Nervous System Tumors; Leukemia; Lymphoma; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: juvenile myelomonocytic leukemia; relapsing chronic myelogenous leukemia; unspecified childhood solid tumor, protocol specific; childhood chronic myelogenous leukemia; childhood acute promyelocytic leukemia (M3); recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; childhood central nervous system germ cell tumor; childhood choroid plexus tumor; childhood craniopharyngioma; childhood infratentorial ependymoma; childhood grade I meningioma; childhood grade II meningioma; childhood grade III meningioma; childhood supratentorial ependymoma; recurrent childhood brain stem glioma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood ependymoma; recurrent childhood medulloblastoma; recurrent childhood supratentorial primitive neuroectodermal tumors; recurrent childhood visual pathway and hypothalamic glioma; recurrent childhood visual pathway glioma; high-grade childhood cerebral astrocytoma; low-grade childhood cerebral astrocytoma; recurrent childhood brain tumor; childhood spinal cord tumor; recurrent/refractory childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; recurrent childhood large cell lymphoma; stage IV childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; stage IV childhood small noncleaved cell lymphoma; childhood grade III lymphomatoid granulomatosis; childhood nasal type extranodal NK/T-cell lymphoma; recurrent childhood grade III lymphomatoid granulomatosis; recurrent childhood pineoblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Leukemia; Lymphoma; Leukemia, Myelomonocytic, Juvenile; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Choroid Plexus Neoplasms; Astrocytoma; Familial ependymoma; Medulloblastoma; Optic Nerve Glioma; Spinal Cord Neoplasms; Recurrence; Dendritic Cell Sarcoma, Interdigitating; Burkitt Lymphoma; Lymphoma, Extranodal NK-T-Cell | interventions — N(alpha)-(4-amino-4-deoxypteroyl)-N(delta)-hemiphthaloyl-L-ornithine; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: talotrexin
Procedure: chemotherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as talotrexin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase I trial is studying the side effects and best dose of talotrexin in treating young patients with recurrent solid tumors or leukemia that is recurrent or does not respond to treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Estimate the maximum tolerated dose (MTD) and recommended phase II dose of talotrexin in younger patients with recurrent solid tumors or recurrent or refractory leukemia.
* Determine the toxicity of this drug in these patients.

Secondary

* Determine the antitumor activity of this drug in these patients.
* Assess the tolerability of the defined MTD of this drug in these patients.

OUTLINE: This is a dose-escalation, multicenter study. Patients are stratified according to diagnosis (solid tumor vs leukemia).

* Stratum 1 (recurrent solid tumor): Patients receive talotrexin IV over 10 minutes on days 1 and 8. Treatment repeats every 21 days for up to 17 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of talotrexin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity (DLT).

* Stratum 2 (recurrent or refractory leukemia): A cohort of 3-6 patients with leukemia receive treatment as in stratum 1 at the MTD determined in stratum 1. If 2 or 3 or 2 of 6 patients experience a DLT at the solid tumor MTD, accrual is stopped.

After completion of study treatment, patients are followed for 30 days.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of either of the following:

  * Recurrent solid tumor

    * Histologically confirmed* malignancy at original diagnosis or relapse
    * Measurable or evaluable disease
    * Lymphoma or primary CNS tumor allowed

      * Patients with CNS tumors must be on a stable or decreasing dose of dexamethasone for the past 7 days
  * Recurrent or refractory leukemia

    * Confirmed relapse, as defined by M3 marrow (25% blasts in bone marrow aspirate or biopsy)
    * Active extramedullary disease allowed provided there is no leptomeningeal involvement NOTE: *Histological confirmation not required for intrinsic brain stem tumors
* Bone marrow metastases allowed

  * Not refractory to red blood cell or platelet transfusion
* No pleural effusion or significant ascites
* No known curative therapy or therapy proven to prolong survival with an acceptable quality of life exists
* No Down syndrome

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) 50-100% (for patients > 10 years of age) OR Lansky PS 50-100% (for patients ≤ 10 years of age)
* Absolute neutrophil count ≥ 1,000/mm³ (for patients with solid tumors without bone marrow involvement)
* Platelet count ≥ 100,000/mm³ (transfusion independent)
* Hemoglobin ≥ 8.0 g/dL
* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min OR creatinine adjusted according to age as follows:

  * No greater than 0.6 mg/dL (1 year to 23 months)
  * No greater than 0.8 mg/dL (2 to 5 years)
  * No greater than 1.0 mg/dL (6 to 9 years)
  * No greater than 1.2 mg/dL (10 to 12 years)
  * No greater than 1.4 mg/dL (13 years and over [female])
  * No greater than 1.5 mg/dL (13 to 15 years [male])
  * No greater than 1.7 mg/dL (16 years and over [male])
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT ≤ 110 U/L (ULN is 45 U/L)
* Albumin ≥ 2 g/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled infection
* No known condition that, in the opinion of the investigator, would preclude study compliance

PRIOR CONCURRENT THERAPY:

* Recovered from all prior treatment-related toxicity
* At least 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosourea) (for patients with solid tumors)
* At least 24 hours since prior cytoreduction therapy initiated with hydroxyurea (for patients with leukemia)
* At least 2 weeks since prior local palliative radiotherapy (small port)
* At least 6 months since prior total-body irradiation (TBI), craniospinal radiotherapy, or ≥ 50% radiotherapy to the pelvis
* At least 6 weeks since prior substantial bone marrow radiotherapy
* At least 3 months since prior stem cell transplant or rescue without TBI

  * No evidence of active graft-versus-host disease
* At least 7 days since prior growth factor therapy
* At least 7 days since prior biological therapy
* No nonsteroidal anti-inflammatory drugs (NSAIDs), aspirin or other salicylates, penicillins, sulfa drugs (bactrim, septra), ciprofloxacin, tetracycline, thiazide diuretics, or probenecid within 2 days prior to, during, or within 5 days after treatment with talotrexin
* No long-acting NSAIDs (e.g., nabumetone, naproxen, oxaprozin, piroxicam) within 5 days prior to, during, or within 5 days after treatment with talotrexin
* No concurrent investigational drugs
* No concurrent anticancer agents or therapy (e.g., chemotherapy, radiotherapy, immunotherapy, or biologic therapy)

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2007-02; Primary Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of talotrexin
Toxicity

SECONDARY OUTCOMES:
Antitumor activity
Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: James Croop, MD, PhD, Study Chair — Riley's Children Cancer Center at Riley Hospital for Children; Sultan Ahmed Pradhan, MD, Study Chair — Tata Memorial Hospital